CLINICAL TRIAL: NCT06668194
Title: A Randomized Clinical Trial Comparing the Effect of Force Magnitude on the Rate of Canine Retraction and Gingival Crevicular Fluid Proteome Profile
Brief Title: Effect of Force Magnitude on Canine Retraction and Gingival Crevicular Fluid Proteome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Charles Burstone Foundation (Unknown)
Responsible Party: Principal Investigator, Flavio Uribe, Professor, UConn Health
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-314-2
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Tooth Crowding
Keywords: Orthodontic space closure; Canine retraction; Gingival crevicular fluid; Proteomics
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: Split mouth design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Light force (150g Niti Coil Spring) (Active Comparator): One of the maxillary canines to be retracted will be assigned to the light force group randomly. Patients' participation in the study (T0) will be started at the stage of canine retraction. At this appointment, 0.019 x 0.025-inch stainless steel archwire will be placed; power arms will be fabricated from 17x25-inch stainless steel on the maxillary first molars and canines. The height of the power arm will be matched with the center of resistance of both canines and molars based on the root length measured on the periapical radiographs. The archwire will be engaged in the canine bracket using stainless steel ligature wire. NiTi coil spring calibrated for force magnitude (150g) at oral temperature will be used to deliver the assigned force will be engaged from the first molars to the canine power arms.
  Interventions: Device: Light Force (150g Niti Coil)
- Heavy force (400g NiTi Coil Spring) (Experimental): One side of the maxillary canines to be retracted will have a heavy force assigned randomly. Patients' participation in the study (T0) will be started at the stage of canine retraction. At this appointment, 0.019 x 0.025-inch stainless steel archwire will be placed; power arms will be fabricated from 17x25-inch stainless steel on the maxillary first molars and canines. The height of the power arm will be matched with the center of resistance of both canines and molars based on the root length measured on the periapical radiographs. The archwire will be engaged in the canine bracket using stainless steel ligature wire. NiTi coil spring calibrated for force magnitude (400g) at oral temperature will be used to deliver the assigned force will be engaged from the first molars to the canine power arms.
  Interventions: Device: Heavy Force (400 g Niti coil)

INTERVENTIONS:
Device: Light Force (150g Niti Coil) — Patients' participation in the study (T0) will be started at the stage of canine retraction. At this appointment, 0.019 x 0.025-inch stainless steel archwire will be placed; power arms will be fabricated from 17x25-inch stainless steel on the maxillary first molars and canines. The height of the power arm will be matched with the center of resistance of both canines and molars based on the root length measured on the periapical radiographs. The archwire will be engaged in the canine bracket using stainless steel ligature wire. NiTi coil spring calibrated for force magnitude (150g) at oral temperature will be used to deliver the assigned force will be engaged from the first molars to the canine power arms
  Arms: Light force (150g Niti Coil Spring)
Device: Heavy Force (400 g Niti coil) — Patients' participation in the study (T0) will be started at the stage of canine retraction. At this appointment, 0.019 x 0.025-inch stainless steel archwire will be placed; power arms will be fabricated from 17x25-inch stainless steel on the maxillary first molars and canines. The height of the power arm will be matched with the center of resistance of both canines and molars based on the root length measured on the periapical radiographs. The archwire will be engaged in the canine bracket using stainless steel ligature wire. NiTi coil spring calibrated for force magnitude (400g) at oral temperature will be used to deliver the assigned force will be engaged from the first molars to the canine power arms
  Arms: Heavy force (400g NiTi Coil Spring)

SUMMARY:
This study aims to examine the effect of force levels in orthodontic treatment during canine retraction. Force levels refer to the pressure applied by the orthodontic devices to move teeth. Data collection will include gingival fluid, dental molds from a digital scanner, and x-rays of the upper canine region on both sides of the mouth during treatment. The null hypothesis to be tested is that there is no significant difference in the rate of canine movement between the light force and the heavy force levels.

DETAILED DESCRIPTION:
Patients' participation in the study at the first visit (T0) Timepoint 0, will be started at the stage of canine retraction. At this appointment, 0.019 x 0.025-inch stainless steel archwire will be placed; power arms will be fabricated from 17x25-inch stainless steel on the maxillary first molars and canines. The height of the power arm will be matched with the center of resistance of both canines and molars based on the root length measured on the periapical radiographs. The archwire will be engaged in the canine bracket using stainless steel ligature wire.

At the T0 appointment, before applying the retraction force, periapical radiographs of canines (with coronal and apical reference wires for calibration and magnification correction) and GCF (gingival crevicular fluid) samples of each canine will be collected. Gingival sulcus of mesial and distal to canine (bilaterally) will be chosen as sites for GCF sample collection. The study coordinator will take a digital scan using iTero® Element™ in the clinic as the baseline (T0). As the split-mouth design will be applied in this study, right and left sides will be assigned randomly for either 150gm (light force) or 400gm force (heavy force) for each subject. NiTi coil spring calibrated for force magnitude at oral temperature will be used to deliver the assigned force will be engaged from the first molars to the canine power arms. IRB-approved written instructions will also be provided to all the participants. Follow-up visits will be scheduled. After applying the force, follow-up visits will be scheduled at (T1) 1-2 weeks, (T2) 4-5 weeks, (T3) 8-9 weeks, (T4)12-13 weeks, and (T5)16-17 weeks. A new digital scan will be taken at each study appointment (T0 - T5). These digital scans will be used for tooth movement measurements. GCF samples (mesial and distal to canines bilaterally) will be collected only for the first 3 appointments (T0 - T2) for the first 10 participants only in this study.

Periapical radiographs for canines on both sides will be obtained on (T0) Timepoint 0, and (T3) 8-9 weeks and (T5) 16-17 weeks of the study for each participant and analyzed to measure the EARR (external apical root resorption). Following the last study visit, all subjects' treatment will continue as recommended by the primary orthodontic care provider. No new data will be reviewed or collected after (T5).

ELIGIBILITY:
Inclusion Criteria:

* Healthy patient, non-smoker
* Age: 11 - 16 years of age, inclusive.
* A full complement of dentition (central incisor to 1st molar) in the four quadrants, except second molars
* Patients requiring at least upper bilaterally maxillary 1st premolar extraction as a treatment plan (Class I bimaxillary protrusion/ crowding or Class II maxillary dentoalveolar protrusion/ crowding)
* At least 5 mm of space left between canine and 2nd premolar to be closed at the time of canine retraction
* At least six months after the extraction of first premolars and in a 0.019 x 0.025-inch stainless steel archwire in the maxilla
* The ability to read and understand English and to provide informed consent

Exclusion Criteria:

* Patients under 11 years of age and over the age of 16.
* Non-extraction treatment plan
* Extraction of maxillary tooth other than first premolars bilaterally.
* Evidence of poor oral hygiene
* Evidence of previous root resorption
* Missing or impacted tooth in any of the quadrant except 3rd molars.
* Medical issues that affect tooth movement
* Inability to provide oral and written consent to participate.
* Patient on medications that may alter bone metabolisms like bisphosphonates, oral contraceptives, or PTH (parathyroid hormone)
* Chronic illness or syndromic patients.
* Pregnant women, prisoners, and decisional impaired

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Male and female
Enrollment: 40 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Canine retraction | 16-17 weeks
  Amount of canine distal displacement in all 3 dimensions with 6 degrees of freedom will be measured through 17 weeks
Gingival crevicular fluid proteomic analysis | 4-5 weeks
  Collected GCF samples from time point (T0, T1 and T2) and same sides (left or right) and aspect of tooth (mesial or distal) from 10 patients for each of the maxillary canines (total of 12 samples per patient). GCF will be collected for the following time points: T0, T1, and T3. A total of 120 samples will be sent for a non-labeled method of proteomic analysis. This will indicate the change in expression of various proteins in GCF samples throughout treatment.

SECONDARY OUTCOMES:
External apical root resorption (EARR) | 16-17 weeks
  The amount of root resorption on the canines as they are being retracted will be measured radiographically before starting retraction, at 8-9 weeks, and at 16-17 weeks.
Maxillary first molar 3 dimensional displacement | 16-17 weeks
  Maxillary first molar displacement in response to a heavy and light force will be characterized in 3D through the 17 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Uribe, DDS, MDentSc, Principal Investigator — UConn Health
Locations (1):
- Department of Orthodontics, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Data on primary and secondary outcomes
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be available approximately 1 year after recruiting the first patient and 1 year after the recruitment of the last patient.
Access Criteria: A data sharing agreement must be signed. The documents should be submitted to the PI by email at furibe@uchc.edu

REFERENCES:
- [Background] Ren Y, Maltha JC, Van 't Hof MA, Kuijpers-Jagtman AM. Optimum force magnitude for orthodontic tooth movement: a mathematic model. Am J Orthod Dentofacial Orthop. 2004 Jan;125(1):71-7. doi: 10.1016/j.ajodo.2003.02.005. PMID 14718882
- [Background] Yee JA, Turk T, Elekdag-Turk S, Cheng LL, Darendeliler MA. Rate of tooth movement under heavy and light continuous orthodontic forces. Am J Orthod Dentofacial Orthop. 2009 Aug;136(2):150.e1-9; discussion 150-1. doi: 10.1016/j.ajodo.2009.03.026. PMID 19651334
- [Background] Iwasaki LR, Liu Y, Liu H, Nickel JC. Speed of human tooth movement in growers and non-growers: Selection of applied stress matters. Orthod Craniofac Res. 2017 Jun;20 Suppl 1:63-67. doi: 10.1111/ocr.12161. PMID 28643922